CLINICAL TRIAL: NCT04507659
Title: A Multi-center, Randomized, Double-blind, Placebo, Parallel-controlled Phase Ⅱ Clinical Trial of Jaktinib Hydrochloride Tablets in the Treatment of Patients With Active Ankylosing Spondylitis
Brief Title: Jaktinib Hydrochloride Tablets In The Treatment of Active Ankylosing Spondylitis
Acronym: AS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Suzhou Zelgen Biopharmaceuticals Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ZGJAK008
Record Dates: First submitted 2020-08-04; First posted 2020-08-11 (Actual); Last update posted 2023-03-29 (Actual); Status verified 2023-03

CONDITIONS: Ankylosing Spondylitis
MeSH Terms: conditions — Spondylitis, Ankylosing

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Jaktinib 100mg (Experimental): 100 mg bid.po
  Interventions: Drug: Jaktinib Hydrochloride Tablets
- Jaktinib 75mg (Experimental): 75 mg bid.po
  Interventions: Drug: Jaktinib Hydrochloride Tablets
- Placebo (Placebo Comparator): Placebo bid.po
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Jaktinib Hydrochloride Tablets — Morning: 2*50mg simulated tablets and 1*75mg Jaktinib Hydrochloride Tablets; Evening: 2*50mg simulated tablets and 1*75mg Jaktinib Hydrochloride Tablets.
  Other Names: Jaktinib
  Arms: Jaktinib 75mg
Drug: Jaktinib Hydrochloride Tablets — Morning: 1*75mg simulated tablet, 2*50mg Jaktinib Hydrochloride Tablets; Evening: 1*75mg simulated tablet, 2*50mg Jaktinib Hydrochloride Tablets.
  Other Names: Jaktinib
  Arms: Jaktinib 100mg
Drug: Placebo — Morning: 1*75mg simulated tablet, 2*50mg simulated tablets; Evening: 1*75mg simulated tablet, 2*50mg simulated tablets.
  Arms: Placebo

SUMMARY:
This trial uses a multi-center, randomized, double-blind, placebo, parallel-controlled design, and it is expected that about 105 cases will be enrolled in about 10 sites.

DETAILED DESCRIPTION:
The study is divided into two stages, the first stage (1-16 weeks) is the main study; the second stage (17-32 weeks) is the extended study. This study set up 3 groups:Jaktinib Hydrochloride Tablets 75mg Bid group, 100mg Bid group and a placebo control group. The subjects were randomly enrolled in the group 1:1:1.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65, both gender;
* Active Ankylosing Spondylitis;
* Participants who have been treated with non-steroidal anti-inflammatory drugs(NSAIDs) and still have active disease, or Participants who are intolerant to NSAIDs and stop the drug;
* Participants receiving low-dose oral glucocorticoid therapy (≤10mg/d prednisone) should maintain a stable medication regimen for at least 4 weeks before the first dose of this study. Do not adjust the dose during the entire study period except in emergency situations.
* Participants receiving other non-prohibited co-drugs should maintain a stable medication regimen for at least 7 days before the first dose of this study;
* Understand and voluntarily signed informed consent.

Exclusion Criteria:

* A history of known or suspected complete spinal rigidity, or clinical and imaging confirmed complete spinal rigidity;
* A history of any other autoimmune rheumatic disease;
* Any history of joint prosthesis infection, and the prosthesis is still in place;
* Participants who are using strong opioid analgesics (such as methadone, hydromorphone, morphine, etc.);
* Participants who have been treated with any JAK inhibitors (such as Tofacitinib, Baricitinib, Ruxolitinib, Filgotinib, Upadacitinib, etc.);
* Participants who have drug abuse or alcohol dependence;
* Participants who have had herpes virus infection in the past month;
* Participants who have a history of venous thrombosis (regardless of current treatment);
* Any significant clinical and laboratory abnormalities that the investigator believes will affect the safety evaluator；
* Participants who cannot be treated and followed up according to the trial protocol;
* Any Participant considered by the investigator to be unsuitable to participate in this clinical study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2022-08-02 (Actual); Study Completion 2022-08-02 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants Achieving 20 Percent (%) Improvement in Assessment of SpondyloArthritis International Society (ASAS) Score (ASAS 20) at Week 16 | Week 16
  ASAS20 responder had improvement of greater than or equal to (≥) 20% and ≥1 unit in at least 3 domains (on a scale of 0 [least] to 10 [worst]) and no worsening of ≥20% and less than or equal to (≤)1 unit in the remaining domain. The domains are: Patient's Global Assessment of Disease Activity, spinal pain, function and inflammation (from Bath Ankylosing Spondylitis Disease Activity Index [BASDAI]). Missing data were handled by nonresponsive (NRI)/ last observation carried forward (LOCF). Missing values due to a subject dropping out from the study were handled by setting the ASAS20 value to NRI. The LOCF approach was applied to missing components, if just some of the components of the ASAS20 were missing.

SECONDARY OUTCOMES:
Percentage of Participants Achieving ASAS 20 at Week 2, 4, 8, 12, 20, 24, and 32 | Week 2,4,8,12,16,20,24,32
  It assess the disease activity. It was evaluated with a 6-question questionnaire. After taking the answer of each question out of 10, the total of the points was calculated by dividing the number of questions.The score range was 0-10, the low score meant that the spinal movement was better.
Percentage of Participants Achieving ASAS 40 at Week 2, 4, 8, 12, 16, 20, 24, and 32 | Week 2,4,8,12,16,20,24,32
  ASAS 40 is defined as ≥40% and absolute change of ≥2 units in at least 3 domains on a 0-10 scale (0=no disease activity, 10=high disease activity), and no worsening in the remaining domain. Missing data were handled by NRI/LOCF.
Percentage of Participants Achieving ASAS 70 at Week 2, 4, 8, 12, 16, 20, 24, and 32 | Week 2,4,8,12,16,20,24,32
  It characterises the spinal mobility of patients with ankylosing spondylitis. Cervical rotation, tragus-wall distance, lateral lumbar flexion, anterior lumbar flexion (modified schober), intermalleolar distance were measured. The score range was 0-10, the low score meant that the spinal movement was better.
Percentage of Participants Achieving ASAS 5/6 Response at Weeks 2, 4, 8, 12, 16, 20, 24, and 32 | Week 2,4,8,12,16,20,24,32
  ASAS5/6 consists of 6 domains: the 4 used in ASAS20 (Patient's Global Assessment of Disease Activity, spinal pain, function, inflammation plus spinal mobility and an acute phase reactant, C Reactive Protein (CRP). ASAS 5/6 is defined as ≥20% improvement in at least 5 domains and no worsening in the remaining domain. Missing data were handled by NRI/LOCF.

CONTACTS AND LOCATIONS:
Overall Officials: Chunde Bao, MD, Principal Investigator — RenJi Hospital
Locations (1):
- Renji Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wang J, Bao C, Dai Q, Xu A, Ye Y. Efficacy and safety of jaktinib hydrochloride tablets in active axial spondyloarthritis: a multicentre, randomised, double-blind, placebo-controlled phase II clinical trial. RMD Open. 2025 Jan 2;11(1):e004865. doi: 10.1136/rmdopen-2024-004865. PMID 39753296